CLINICAL TRIAL: NCT02517411
Title: Effects of a Physiotherapy Program in Patients With Stable Chronic Obstructive Pulmonary Disease
Brief Title: Physiotherapy in Patients With Stable Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, PhD, Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DF0058UG
Record Dates: First submitted 2015-08-02; First posted 2015-08-07 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: COPD
Keywords: COPD; physiotherapy; Stable disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Standard of Care; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): COPD patients with stable disease will be recruited and they will receive physiotherapy added to standard care.
  Interventions: Other: Physiotherapy added to standard care
- Control group (Other): COPD patients with stable disease will be recruited and they will receive standard care.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Standard care — The standard care of stable COPD is based on long-acting bronchodilators (LABD).
  Other Names: standard treatment
  Arms: Control group
Other: Physiotherapy added to standard care — The treatment will be based on domiciliary physiotherapy program during 8 weeks, twice a week added to standard care. The duration of the sessions will be 45-60 minutes. The physiotherapy treatment includes: breathing exercises, electrostimulation in quadriceps with voluntary contraction and exercises with theraband. This will be a home-based program supervised by a physiotherapist.
  Other Names: Physiotherapy; Home-based program; Domiciliary physiotherapy
  Arms: Experimental group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a lung disease that is characterized by incompletely reversible airflow obstruction. It is projected to be the fifth leading burden of disease worldwide by the year 2020. Pulmonary dysfunction reduces exercise capacity in COPD patients, and it has been previously shown that COPD patients suffer deterioration in their quality of life. The objective of this study is to examine the effects of a physical therapy intervention in stable patients with COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is one of the leading diseases causing mortality and morbidity, despite advanced pharmacotherapy and therapeutic management. Although COPD primarily affects the lungs, it also implies extrapulmonary manifestations, such as nutritional depletion, skeletal muscle dysfunction, and abnormal respiratory muscles.

Pulmonary rehabilitation is widely used to treat COPD patients and it has been shown that pulmonary rehabilitation should be implemented at all COPD stages, bringing them benefits in terms of improved exercise capacity, symptoms, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis
* No contraindication of physiotherapy.
* Signed written consent.
* Medical approval for inclusion.

Exclusion Criteria:

* Acute exacerbation in the previous month
* Contraindications of physiotherapy.
* Neurological, orthopedic or heart disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Changes in Muscle strength | Baseline, 8 weeks
  Quadriceps strength will be assessed with a portable dynamometer.
Changes in Exercise capacity | Baseline, 8 weeks
  Five times sit to stand test (5STS) will be used to assess exercise capacity, 5STS is a simple assessment tool that is feasible in all healthcare settings, and may be a rapid method of assessing changes in exercise capacity in COPD and screening for poor physical functioning individuals.

SECONDARY OUTCOMES:
Changes in Respiratory function | Baseline, 8 weeks
  Spirometry is regarded as the gold standard measure of respiratory function. Spirometry will be performed according to the American Thoracic Society (ATS) criteria.
Changes in Dyspnea perception | Baseline, 8 weeks
  Dyspnea perception will be assessed with Borg modified scale. Patients will classify their breathlessness between 0 and 10.
Changes in Quality of life | Baseline, 8 weeks
  EuroQol-5D (EQ-5D) will be used to assess quality of life. EQ-5D is a generic questionnaire and consists of two parts, the EQ-5D Visual analogue scale (VAS) and the EQ-5D index. The EQ-5D VAS consists on a vertical rating scale from 0 to 100 (0 = death/worst possible health state and 100 = best possible health state). The EQ-5D index is a five-item questionnaire (mobility, self-care, usual activity, pain/discomfort and anxiety/depression).
Changes in Fatigue | Baseline, 8 weeks
  Fatigue will be assessed with the Fatigue Severity Scale (FSS). The FSS is a nine-item instrument designed to assess fatigue as a symptom of a variety of different chronic conditions and disorders. The scale addresses fatigue's effects on daily functioning, querying its relationship to motivation, physical activity, work, family, and social life, and asking respondents to rate the ease with which they are fatigued and the degree to which the symptom poses a problem for them.
Impact of COPD | Baseline, 8 weeks
  The impact of COPD in patient's life will be evaluated with COPD Assessment Test (CAT) that is a simple instrument to quantify chronic obstructive pulmonary disease (COPD) impact in routine practice.

OTHER OUTCOMES:
Quality of life related to respiratory symptoms | Baseline
  Saint George Respiratory Questionnaire (SGRQ) will be also used to evaluate the quality of life of patients in the previous year. It includes 50 items, divided into three domains: Symptoms, Activity and Impacts. A score is calculated for each domain and a total score including all items is also obtained. Low scores indicate better health related quality of life.
Peripheral vascular status | Baseline
  Ankle-brachial index will be used to predict the presence or absence of peripheral arterial disease.
Physical activity | Baseline
  Modified Baecke Questionnaire will be used to assess the physical activity levels. It is a frequently used questionnaire to measure habitual physical activity in the elderly.
Cognitive status | Baseline
  Cognitive status will be assessed with Montreal Cognitive Assessment test (MoCA) which is a cognitive screening test designed to assist Health Professionals for detection of mild cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Department of Physical Therapy, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided